CLINICAL TRIAL: NCT03460847
Title: Can Fecal Microbiota Alterations Predict a Refractory Disease Course to Standard Steroid Therapy in Patients With Active Ulcerative Colitis?
Brief Title: Fecal Microbiota Alterations in Steroid Refractory Active Colitis Ulcerosa
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-316 ex 16/17
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Steroids — Patients with active colitis ulcerosa who need steroids because of their disease course. 1mg/kg bodyweight for one week, followed by a tapping periode.
  Other Names: Aprednisolon, Prednisolut

SUMMARY:
Alterations in the intestinal microbiota have been associated to disease pathogenesis in ulcerative colitis. Refractory disease to standard medical therapy as corticosteroids often leads to an unfavourable course in patients suffering from this disorder. This study proposal aims at investigating changes in the intestinal microbiota that can predict a therapy refractory course of ulcerative colitis (UC) and may be used to identify high risk patients in an early phase of their disease.

DETAILED DESCRIPTION:
The Investigators suggest that certain alterations in the intestinal microbiota are at least in part responsible for the inability of some patients to response to steroid therapy and probably also for the failure to other immunosuppressive therapies. Certain pathobionts have the capability to stimulate the mucosal immune system, thereby leading to chronic inflammation. On the other hand, commensals are necessary for repair processes in the mucosa and are providing metabolites that are used as an energy source for the colonic epithelium. An increase in pathobionts in combination with a lack of certain commensals might therefore maintain colonic inflammation despite immunosuppressive therapy with systemic steroids in patients with UC.

The investigators therefore plan to investigate the intestinal microbiota in UC patients before and 4 weeks after a systemic corticosteroid therapy and correlate potential alterations of the microbiota to the therapeutic response. Other factors like concomitant UC treatment, disease severity, disease extent and environmental factors will also be correlated to changes in the microbiota.

In the subgroup of patients not responding to steroids and requiring a rescue therapy with infliximab or a calcineurin Inhibitor, the predictive value of microbiota alterations will also be investigated.

If certain bacterial taxa can predict a steroid refractory and an unfavorable disease course, the results of this study will help in identifying possible microbiota based biomarkers for an individualized treatment approach in UC patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis with a Lichtiger score ≥4
* Patient scheduled for steroid therapy with systemic steroids (prednisolone or methylprednisolone) at standard dosing and patients who started steroid therapy not longer than 48 hours prior to the study inclusion.
* Written informed consent
* Established or suspected diagnosis of ulcerative colitis or indeterminate colitis

Exclusion Criteria:

* No follow up possible
* Bacterial intestinal infections (C. difficile, Salmonella, EHEC, Campylobacter, Shigella, Yersinia), parasitic or viral infection causing acute infectious diarrhea at baseline.
* Diagnosis of Crohn´s disease
* Planned initiation or discontinuation of probiotic therapy between baseline and follow up visit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from an active colitis ulcerosa and requiring steroids as therapy.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Microbiota alterations | 28 days
  To assess if alterations of the fecal microbiota are associated with a failure to respond to steroid therapy within 28 days in patients with ulcerative colitis. The microbiota will be assessed by 16s RNA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hoegenauer, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- LKH Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided